CLINICAL TRIAL: NCT01722630
Title: Dopamine Infusion and Crystalloids Administration Improve Renal Function During Laparoscopic Surgery
Brief Title: Renal Function During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesca Bevilacqua, Medical Doctor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRF-2012-DH
Record Dates: First submitted 2012-11-02; First posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Intra Operative Fluid Management
Keywords: dopamine; laparoscopy; fluid management
MeSH Terms: interventions — Dopamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): Patients received intravenously saline solution at 5 ml/Kg/h
- dopamine (Experimental): Patients received intravenously saline solution at 5 ml/Kg/h and dopamine at 3 mcg/Kg/min
  Interventions: Drug: Dopamine
- crystalloids (No Intervention): Patients received intravenously saline solution at 10 ml/Kg/h

INTERVENTIONS:
Drug: Dopamine
  Other Names: Revivan
  Arms: dopamine

SUMMARY:
Aim of this study was to investigate the cardiac and renal responses to the administration of different amount of crystalloids, with and without dopamine, during gynaecological laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I
* age 24-42
* patients undergoing gynaecological laparoscopy

Exclusion Criteria:

* cardiovascular diseases
* renal and endocrine disorders
* obesity (BMI > 30 Kg/m2)
* the assumption of drugs that could interfere with renal parameters considered in the study

Ages: 24 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
estimated glomerular filtration rate, tissue Doppler imaging, E/Ea | patients will be followed for the duration of surgery, an expected average of 3 hours
  EGFr, tissue Doppler imaging and E/Ea are registered after the induction of pneumoperitoneum and Trendelemburg position, and compared to those registered before the induction of anesthesia.

SECONDARY OUTCOMES:
total intra operative diuresis (TID) | patients will be followed for the duration of surgery, an expected average of 3 hours
  TID will be measured at the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the sacred Heart, Rome, Rome, Italy